CLINICAL TRIAL: NCT06722625
Title: Telemedical Care System for the Treatment of Arterial Hypertension Using Recommendation Algorithms to Support Diagnostic and Therapeutic Decisions
Brief Title: Telemedical Algorithm-Supported Care for Hypertension
Acronym: SOT-ART-HT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2/XXI/2023
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Arterial Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Standard care involving regular visits to a hypertension clinic. Patients in the control group will receive standard care. They will have appointments according to the guidelines of the Polish Society of Hypertension -initially once a month and, after achieving control (i.e., blood pressure in office measurement < 140/90 mmHg), once every 3 months.
- Study group (Experimental): In the intervention group, a care model using a system implementing an algorithm that supports therapeutic and diagnostic decisions made by the doctor in the care of patients with AH will be applied. The algorithm identifies patients who have or have not achieved therapeutic goals and suggests actions for specific patients, but the final therapeutic and diagnostic decisions are always made by the doctor. It is emphasized that the treating physician is not bound by the algorithm's recommendations.
  Interventions: Other: Evaluation of a blood pressure monitoring system with an integrated algorithm that supports the doctor's decision-making process

INTERVENTIONS:
Other: Evaluation of a blood pressure monitoring system with an integrated algorithm that supports the doctor's decision-making process — Receiving remote care facilitated by a specialized informatic system to support the physician
  Arms: Study group

SUMMARY:
Hypertension is a major global health issue, affecting around 9 million people in Poland. While some studies indicate that telemonitoring benefits patients with hypertension, there is a lack of research evaluating tools that assist doctors in managing these patients. The objective of this study is to assess a blood pressure monitoring system with an integrated algorithm that aids doctors in the decision-making process.

DETAILED DESCRIPTION:
The SOT-ART-HT study is a single-center, randomized, open-label trial aimed at comparing two strategies for managing arterial hypertension. Patients in the control group will receive standard care, which includes regular visits to a hypertension clinic, while those in the intervention group will receive remote care through a specialized tele-informatic system designed to assist the physician. The trial will involve 200 participants, aged 18-80, with confirmed arterial hypertension and uncontrolled office blood pressure at the screening visit. Both primary and secondary outcomes will be evaluated, with the study expected to be completed after 2026. However, early termination could occur if required by regulatory bodies, an Ethics Committee, or the Scientific Research Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signing an informed consent to participate in the study.
2. Age between 18 and 80 years.
3. Diagnosis of hypertension according to the Polish Society of Hypertension criteria from 2019, either already treated or newly diagnosed.
4. Blood pressure exceeding 140/90 mmHg in office measurements (during the screening visit).

Exclusion Criteria:

1. Suspicion or diagnosis of secondary hypertension.
2. Pregnant women, breastfeeding women, or those planning pregnancy during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Achieving Arterial Blood Pressure Control | After completing the presumed six-month follow-up of the last participant
  Time from study initiation to the day of achieving arterial blood pressure control, defined as a 7-day mean of home blood pressure measurements below 135/85 mmHg
Assessment of Achieving Arterial Blood Pressure control at 6 months | After 6 months of participating
  The time from study initiation to 6 months of participation, achieving arterial blood pressure control, defined as a 7-day average of home blood pressure measurements below 135/85 mmHg

SECONDARY OUTCOMES:
Assessment of blood pressure values in 24-hour monitoring, home measurements, and office measurements | Baseline up to approximately six-months of observation
  Analysis of Blood Pressure Values: 24-Hour Monitoring, Home Measurements, and Office Measurements
Assessment of the number of the medical visits | After completing the presumed six-month follow-up of the last participant
  The number of medical visits from study initiation to completion
Assessment of the maintaining blood pressure control | After completing the presumed six-month follow-up of the last participant
  Total time maintaining blood pressure control, defined as the number of days with a 7-day mean of home measurements below 135/85 mmHg
Assessment of the cost of visits | After completing the presumed six-month follow-up of the last participant
  Cost of visits incurred by the medical institution and the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hypertensiology, Angiology and Internal Medicine, Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lipski D, Lewandowska K, Zurek S, Wisniewicz M, Pirog P, Tykarski A, Uruski P. Telemedical care system for the treatment of arterial hypertension using recommendation algorithms to support diagnostic and therapeutic decisions-study protocol for a single-center, randomized, controlled, open-label SOT-ART-HT trial. Trials. 2025 Sep 1;26(1):330. doi: 10.1186/s13063-025-09044-w. PMID 40890870